CLINICAL TRIAL: NCT06998082
Title: A Large Language Model-Driven Multimodal Early Warning Platform for Perioperative Complications in Acute Hemorrhagic Cerebrovascular Disease
Brief Title: AI-Driven Early Warning System for Perioperative Risks in Acute Hemorrhagic Stroke
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yuming Peng, Deputy chief of Department of Anesthesiology, Beijing Tiantan Hospital
Other Study IDs: 20250401
Record Dates: First submitted 2025-05-09; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-04

CONDITIONS: Acute Hemorrhagic Stroke
Keywords: Perioperative Complications; Artificial intelligence in Medicine; Acute hemorrhagic stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with acute hemorrhagic cerebrovascular disease

SUMMARY:
Acute hemorrhagic cerebrovascular disease is a life-threatening condition characterized by sudden onset, rapid progression, multiple complications, poor prognosis, and high mortality. It presents a significant public health burden. During surgical interventions, precise risk stratification and effective perioperative management are crucial to mitigating intraoperative and postoperative complications, optimizing disease diagnosis, guiding severity assessment, and refining anesthesia strategies. Continuous real-time evaluation and dynamic perioperative adjustments are essential to minimize the influence of institutional variability and individual clinician-dependent decision-making. By harnessing big data-driven, evidence-based medical approaches, clinicians can enhance diagnostic accuracy and therapeutic precision, addressing a critical challenge in reducing morbidity and mortality in this patient population.

This study aims to develop a comprehensive multimodal perioperative database and leverage large language models (LLMs) for the efficient extraction of structured demographic and clinical data throughout the perioperative course. By integrating real-time hemodynamic monitoring parameters, the investigators seek to elucidate the relationship between perioperative hemodynamic patterns and the incidence of postoperative complications affecting major organ systems, including the brain, heart, kidneys, and lungs. The ultimate goal is to construct a multimodal fusion early-warning model capable of real-time, simultaneous prediction of multiple perioperative complications. This AI-driven platform will function as a risk stratification and alert system for organ-specific perioperative complications in patients with acute hemorrhagic cerebrovascular disease. By providing evidence-based insights for optimized perioperative management-encompassing early warning mechanisms, diagnostic support, and individualized therapeutic strategies-the system aims to improve clinical outcomes, reduce perioperative morbidity, and lower overall mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 80 years.
* Diagnosis confirmed by preoperative imaging (CT or MRI) of one of the following conditions:
* Intracranial aneurysm
* Arteriovenous malformation (AVM)
* Hemorrhagic moyamoya disease
* Cavernous malformation
* Spontaneous intracerebral hemorrhage
* Undergoing surgery within seven days of symptom onset.

Exclusion Criteria:

* Patients who decline to provide informed consent.
* Patients enrolled in conflicting clinical studies.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators plan to recruit patients aged 18-80 years with acute hemorrhagic cerebrovascular disease from a minimum of three tertiary Grade A general hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 1533 (Estimated)
Dates: Start 2025-07-06 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measures were postoperative complications involving the neurological, cardiac, pulmonary, and renal systems in patients with acute hemorrhagic cerebrovascular disease following surgical interventions. | Within 30 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided